CLINICAL TRIAL: NCT06569797
Title: The Effect of Adding Milk Oligosaccharides and Optimizing Multiple Nutrients to Infant Formula on the Growth and Development of Infants Aged 0-1 Years: a Multicenter, Double-blind, Randomized, Controlled Trial
Brief Title: Effect of Oligosaccharides and Optimizing Multiple Nutrients to Infant Formula on Growth and Development of Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heilongjiang Feihe Dairy Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Nan Yi Da Lun (2023) No. 524
Record Dates: First submitted 2024-08-07; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Milk oligosaccharides; multiple nutrients; infants
MeSH Terms: interventions — Oligosaccharides; Lactation

STUDY DESIGN:
Intervention Model Description: multicenter, double-blind, randomized, controlled trial
Who Masked: Participant, Investigator
Masking Description: This clinical study is a double-blind trial, and before unblinding, neither the researchers nor the subjects know whether they belong to the experimental group or the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group (Experimental): Feeding infant formula with added milk oligosaccharides and optimized for multiple nutrients
  Interventions: Dietary Supplement: oligosaccharides and multiple nutrients
- control group (Active Comparator): Feeding with regular infant formula milk powder
  Interventions: Dietary Supplement: no oligosaccharides and optimizing multiple nutrients
- Breastfeeding group (Active Comparator): Breastfeeding with breast milk
  Interventions: Dietary Supplement: breastfeeding

INTERVENTIONS:
Dietary Supplement: oligosaccharides and multiple nutrients — The effect of adding milk oligosaccharides and optimizing multiple nutrients to infant formula on the growth and development of infants aged 0-1 years
  Arms: experimental group
Dietary Supplement: no oligosaccharides and optimizing multiple nutrients — The effect of traditional infant formula milk powder optimized without adding milk oligosaccharides and multiple nutrients on the growth and development of infants aged 0-1 years old.
  Arms: control group
Dietary Supplement: breastfeeding — The impact of breastfeeding on the growth and development of infants aged 0-1 years old.
  Arms: Breastfeeding group

SUMMARY:
The research objective is to compare the effects of infant formula supplemented with milk oligosaccharides and optimized with multiple nutrients on the immune function of infants under 1 year old with conventional infant formula, and to compare the effects of different infant formulas on infant intestinal health, immune function, growth and development, cognitive development, and tolerance with those of breastfed infants.

DETAILED DESCRIPTION:
In this clinical trial, the effects of adding oligosaccharides to breast milk and optimizing multiple nutrients in infant formula, conventional infant formula, and breast milk on the growth and development of infants under 1 year old were evaluated by comparing the intestinal indicators (16s rRNA, SCFAs), inflammatory indicators, nutritional indicators, immune indicators, growth and development indicators, bone development indicators, tolerance indicators, cognitive development, adverse events, and serious adverse events of 80 experimental groups, 80 control groups, and 80 breastfeeding groups

ELIGIBILITY:
Inclusion Criteria:

* 0-28 days after birth;
* Single birth;
* The gestational age is between 37 and 42 weeks;
* Birth weight ranges from 2500 to 4000 grams;
* Parents or guardians agree not to allow infants to participate in other interventional clinical studies during the study period

Exclusion Criteria:

* Artificial assisted reproduction;
* The mother suffers from a disease that may endanger intrauterine growth;
* The mother suffers from pregnancy diabetes or serious metabolic disease or chronic disease during pregnancy
* Suffering from congenital malformations and genetic diseases, chronic diseases, and congenital diseases that may interfere with the investigation;
* Suffering from IgE mediated milk protein allergy, or having factors that increase the risk of milk protein allergy;
* Suffering from acute infection or gastroenteritis;
* Suffering from functional gastrointestinal diseases, such as gastroparesis;
* Currently participating in other clinical trials;
* Researchers cannot determine whether parents have the willingness or ability to comply with the requirements of the protocol.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Intestinal indicators | day 28,180,360
  16s rRNA
Intestinal indicators | day 28,180,360
  SCFAs

SECONDARY OUTCOMES:
Inflammatory markers | day 180,360
  serum hsCRP
Nutritional indicators | day 180,360
  serum albumin
Immune indicators | day 28,180,360
  fecal sIgA
Immune indicators | day 180,360
  blood lymphocyte subsets
Growth and development indicators | day 28,90,180,360
  height
Growth and development indicators | day 28,90,180,360
  weight
Growth and development indicators | day 28,90,180,360
  head circumference
Growth and development indicators | day 28,90,180,360
  chest circumference
Bone development indicators | day 180,360
  osteocalcin
Bone development indicators | day 180,360
  alkaline phosphatase
Tolerance indicators | day 28,90,180,360
  investigation of infant gastrointestinal comfort：In the past week, the average daily number of reflux .The minimum number is 0, and there is no limit to the maximum number.
Tolerance indicators | day 28,90,180,360
  investigation of infant gastrointestinal comfort：In the past week, abdominal pain VAS score of the infant.The minimum score is 0, and the maximum score is 10.
Tolerance indicators | day 28,90,180,360
  investigation of infant sleep crying：In the past week, the average daily crying time.The minimum time is 0 hours and the maximum time is 24 hours.
Tolerance indicators | day 28,90,180,360
  investigation of infant sleep crying：In the past week, the average daily crying frequency.The minimum number of times is 0, and the maximum number of times is unlimited.
Tolerance indicators | day 28,90,180,360
  investigation of infant sleep crying：In the past week, the average daily crying severity. The severity of crying is divided into no crying, mild crying, moderate crying, very crying, and extreme crying.
Tolerance indicators | day 28,90,180,360
  investigation of infant sleep crying：In the past week, the average daily crying daytime and nighttime sleep duration. The minimum time is 0 hours and the maximum time is 12 hours.
Tolerance indicators | day 28,90,180,360
  investigation of infant sleep crying：In the past week, sleep problems of infants.Sleep problems are divided into no problem, minor problem, moderate problem, major problem, and extreme problem.
Tolerance indicators | day 28,90,180,360
  investigation of infant diarrhea and upper respiratory tract infections：The severity of diarrhea and upper respiratory tract infections (colds) in infants from birth until now. The severity level is classified as no problem, minor problem, moderate problem, major problem, and maximum problem.
Tolerance indicators | day 28,90,180,360
  Bristol stool classification of infant feces
Cognitive Development | day 28,90,180,360
  Bailey Infant Development Scale (Version IV) Score（130 or above, very excellent; 120-129, excellent; 110~119, upper middle; 90-109, moderate; 80-89, below average; 70-79, critical state; Below 69, developmental delay）
Cognitive Development | day 180,360
  Serum Amino Acids

OTHER OUTCOMES:
adverse event | 1 year
  adverse event
Serious adverse events | 1 year
  Serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xu Z Wang, doctor, Study Chair — Nanjing Medical University
Locations (1):
- The Seventh Medical Center of the General Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT06569797/Prot_000.pdf